CLINICAL TRIAL: NCT05643287
Title: The Effect of Time on the Outcome of Periodontal Treatment.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 251 Hellenic Air Force & VA General Hospital (Other)
Responsible Party: Principal Investigator, Georgia Malamoudi, Attendant at Periodontology Department of 251 Hellenic Air Force & VA Hospital, 251 Hellenic Air Force & VA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 251Hellenic
Record Dates: First submitted 2022-11-28; First posted 2022-12-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis
Keywords: Periodontitis; Re-evaluation; Non-surgical periodontal treatment
MeSH Terms: conditions — Periodontitis | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontitis patients (Experimental): Periodontitis patients receiving non-surgical periodontal treatment.
  Interventions: Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: Periodontal treatment — Non-surgical periodontal treatment

SUMMARY:
Re-evaluation after non-surgical periodontal treatment remains an integral part of comprehensive periodontal therapy. This re-evaluation determines if a patient is in need either of surgical periodontal therapy or a personalized program of supportive periodontal treatment. However important, this time point is yet to be determined.This interventional study aims to clarify which is the best time to re-evaluate the therapeutic result after non-surgical periodontal treatment.

DETAILED DESCRIPTION:
This randomized clinical trial aims to clarify which is the best time to re-evaluate the therapeutic result after non-surgical periodontal treatment. For this purpose the participants will be recruited among people who come to the Periodontal Department of 251 Hellenic Air Force Hospital for periodontal treatment. Each participant is going to submit informed consent in order to be included in the study. Patients with the diagnosis of Periodontitis will be submitted to non-surgical periodontal treatment with ultrasonic and manual scalers within two sessions, under local anaesthesia. The result of the treatment is going to be evaluated at 6, 12 and 24 weeks after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Systematically healthy adults
* Informed consent form completion
* Periodontitis Diagnosis
* Patients not having received periodontal treatment since 12 months before

Exclusion Criteria:

* Medical History that interferes with wound healing
* Antibiotic and anti-inflammatory drugs intake
* Medication that induces gingival enlargement
* Pregnancy/ Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket Depth 0 | Baseline
  The distance between the gingival margin and the base of the sulcus/pocket
Probing Pocket Depth 1 | 6 weeks after periodontal treatment
  The distance between the gingival margin and the base of the sulcus/pocket
Probing Pocket Depth 2 | 12 weeks after periodontal treatment
  The distance between the gingival margin and the base of the sulcus/pocket
Probing Pocket Depth 3 | 24 weeks after periodontal treatment
  The distance between the gingival margin and the base of the sulcus/pocket

SECONDARY OUTCOMES:
Clinical attachment level | Baseline, 6, 12, 24 weeks after treatment
  The distance between cementoenamel junction and the base of the sulcus/pocket
Plaque Index | Baseline, 6, 12, 24 weeks after treatment
  Number of sites with presence of dental plaque/ total number of sites
Bleeding on Probing | Baseline, 6, 12, 24 weeks after treatment
  Number of sites with presence of bleeding/total number of sites
Tooth Mobility | Baseline, 6, 12, 24 weeks after treatment
  degree of tooth mobility
Furcation involvement | Baseline, 6, 12, 24 weeks after treatment
  Presence or absence of furcation involvement and degree of furcation defect
matrix metalloproteinase | Baseline, 6, 12, 24 weeks after treatment
  matrix metalloproteinase 8 levels in whole saliva
Oral Health Impact Profile (OHIP)-14 Questionnaire | Baseline, 6, 12, 24 weeks after treatment
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: George Koukos, DDS, PhD, Study Director — 251 Hellenic Air Force & VA Hospital

IPD SHARING:
Plan to Share IPD: No